CLINICAL TRIAL: NCT02507401
Title: Mixed-species Biofilm Composition as a Predictor of Device Longevity in Patients Using Silicone Medical Devices
Brief Title: Mixed-species Biofilms and Silicone Device Longevity
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, Alex Brand, Dr, University of Aberdeen
Other Study IDs: 02/035/15
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Total Laryngectomy Patients Who Use Voice Prostheses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Microbes isolated from in-dwelling medical device (voice prostheses) and oral rinse. No patient biomaterial will be collected or retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total laryngectomy patients: Users of voice prostheses

SUMMARY:
The purpose of this study is to determine whether the mix of microbial species isolated from biofilm-clogged voice prostheses is specific to each participant, whether the microbes are orally-derived and whether the presence of specific species is a predictor of the frequency with which patients discard devices due to malfunction. The microbes isolated from discarded devices will be used to test the antimicrobial properties of newly-developed medical silicones.

DETAILED DESCRIPTION:
This study has three primary objectives and one secondary objective:

Primary Objectives

* To understand variation in the composition of mixed-species biofilms on voice prostheses, both between patients and over time within patients. This will enable us to target resistance to specific microbes using chemistry-based approaches in the design of new medical silicones and develop realistic in vitro models using relevant clinical isolates with which to test them.
* To explore the association between the incidence of specific microbes in biofilms, patient factors (use of antimicrobials, antacids and dentures), and increased device-replacement frequency.
* To explore whether the colonising microbes originate from the participants's oral flora.

Secondary Objective

• To study the interactions that occur within the social group of microbes isolated from each voice prosthesis to learn a) whether these species are interdependent, b) whether they cooperate with each other in order to build biofilms and b) which species produce compounds that physically degrade medical polymers.

STUDY DESIGN

Four hypotheses will be addressed by this study:

1. There is a correlation between the presence of certain microbes, or mixes of microbes, and the frequency of device replacement;
2. The source of the problem microbes is the participants's oral flora;
3. Participant-related factors such as continuous exposure of the microbes to antimicrobial or antacid treatments, or the use of dentures, may alter the composition of device biofilms.
4. Identification of problem microbes may assist in the development of new medical silicones that are specifically designed to resist these species.

These hypotheses will be addressed by collection of discarded devices from participants who are users of voice prostheses and registered at the Speech and Voice Clinic, Aberdeen Royal Infirmary (up to 27 people). Participants will be requested to donate discarded devices, mouthwash samples and simple data on recent antimicrobial or antacid treatments, and the use of dentures. The microbes colonising prostheses and contained within mouthwash samples will be isolated and identified and the association between microbial species and patient data over time will be analysed. Microbes will be stored as clinical isolates and used to test biofilm establishment and maintenance on silicones with modified surfaces designed to reduce biofouling.

ELIGIBILITY:
Inclusion Criteria:

* Total larygectomy patients.
* Must be registered at Speech and Voice Clinic, Aberdeen Royal Infirmary

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Users of voice prostheses who are registered at the Speech and Voice Clinic, Aberdeen Royal Infirmary.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Number of microbial species colonising medical device by patient | 12 months
  Quantification of the number of microbial species colonising medical device by patient

SECONDARY OUTCOMES:
Evidence that oral carriage of a specific microbial species constitutes a risk factor for increased frequency of voice prosthesis malfunction | 12 months
  Association of specific organism carriage and frequency of device change.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Brand, BSc PhD, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data are available to the study